CLINICAL TRIAL: NCT02574806
Title: Normal Values of Brain Natriuretic Peptide in Healthy Newborn
Status: Completed | Type: Observational
Sponsor: Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud (Other)
Responsible Party: Sponsor
Other Study IDs: EBNPRNS01
Record Dates: First submitted 2015-10-07; First posted 2015-10-14 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Reference Values of BNP in Healthy Newborn
Keywords: BNP; Reference values; Newborn; Ventricular function; Stress; Pediatrics; Biomarkers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy newborn: Healthy newborn at term of healthy mother.
  Interventions: Procedure: Blood sample and BNP measurement
- Preeclamptic newborn: Newborn at term of mother with pre-eclampsia with severity features.
  Interventions: Procedure: Blood sample and BNP measurement

INTERVENTIONS:
Procedure: Blood sample and BNP measurement — Blood sample of umbilical artery from umbilical cord immediately after birth.

SUMMARY:
Brain natriuretic peptide (BNP) is an important tool for diagnosis, risk stratification and prognosis in pediatric patients with heart failure1. In newborn, after delivery, the BNP plays an important role in cardiopulmonary hemodynamics by stimulating vasodilatation and diuresis. The gradual decrease in pulmonary pressure and the initiation of diuresis as expression of renal maturity could explain the subsequent decrease in serum values. This would suggest that, in healthy newborns, BNP values should be found within a given ranges. However, the evidence suggests an important variability in BNP values 2 - 4. In the other hand, in the newborn with respiratory distress BNP could have a high negative predictive value to rule out acute myocardial processes, as responsible for clinical deterioration, from infectious, metabolic or respiratory processes; with a potential of improvement in medical care. Even the increased use of this biomarker in clinical practice, until our knowledge, BNP normal values remain unknown in the healthy newborn. Therefore, the investigators performed a pioneer study to establish normal values in healthy newborn population. Multi-center, prospective and observational study was carried out. Objective: To establish normal BNP values in healthy newborn.

ELIGIBILITY:
Inclusion Criteria:

* healthy mother with pregnancy at term (38 to 42 gestational weeks) with adequate prenatal care.
* newborns with Apgar score ≥ 7 at 0 and 5 minutes respectively.

Exclusion Criteria:

* newborns of mothers with pregnancy-associated diseases.
* newborns with chromosomopathies detected during the antenatal care and newborns with signs of cardiac and/or respiratory compromise.

Max Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term newborn obtained by vaginal delivery and/or cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
BNP values | within the first minute after birth and data will present through study completion

REFERENCES:
- [Derived] Rodriguez D, Garcia-Rivas G, Laresgoiti-Servitje E, Yanez J, Torre-Amione G, Jerjes-Sanchez C. B-type natriuretic peptide reference interval of newborns from healthy and pre-eclamptic women: a prospective, multicentre, cross-sectional study. BMJ Open. 2018 Oct 17;8(10):e022562. doi: 10.1136/bmjopen-2018-022562. PMID 30337314
- See also: B-type natriuretic peptide reference interval of newborns from healthy and pre-eclamptic women: a prospective, multicentre, cross-sectional study — https://bmjopen.bmj.com/content/8/10/e022562